CLINICAL TRIAL: NCT01107743
Title: Caduet® Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Amlodipine/Atorvastatin (Caduet®) Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A3841063
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Angina Pectoris; Hypercholesterolemia; Familial Hypercholesterolemia
Keywords: Hypertension; Angina pectoris; Hypercholesterolemia; Familial hypercholesterolemia; Japanese; caduet; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Hypertension; Angina Pectoris; Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — amlodipine, atorvastatin drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Amlodipine and Atorvastatin Combination Tablet: Subjects taking Amlodipine and Atorvastatin Combination Tablets
  Interventions: Drug: Amlodipine/Atorvastatin

INTERVENTIONS:
Drug: Amlodipine/Atorvastatin — Amlodipine and Atorvastatin combination Tablet is indicated in following subjects for whom treatment with both amlodipine and atorvastatin is appropriate.
  Subjects with concurrent hypertension or angina pectoris and hypercholesterolemia or familial hypercholesterolemia Indications for amlodipine and atorvastatin.
  For oral use, amlodipine and atorvastatin combination tablet is given once daily. Dosage must be individualized based on dosage and administration for each individual component.
  Amlodipine
  * Hypertension Usual adult dosage is 2.5-5 mg of amlodipine given orally as a single daily dose.
  * Angina pectoris For oral use, the usual adult dosage is 5 mg of amlodipine once daily. Atorvastatin
  * Hypercholesterolemia For oral use, the usual adult dosage is 10-20 mg of atorvastatin once daily.
  * Familial hypercholesterolemia For oral use, the usual adult dosage is 10-40 mg of atorvastatin once daily.
  Other Names: Caduet

SUMMARY:
In this survey, to collect the safety and efficacy information of Amlodipine /Atorvastatin (Caduet® Combination Tablets) in daily medical practice will be examined. In addition, the necessity of special Investigation and post-marketing clinical studies will be examined, while investigating unexpected adverse drug reactions during the survey period and understanding of the status of frequency of adverse drug reactions in daily medical practice.

DETAILED DESCRIPTION:
All the subjects whom an investigator prescribes the first Amlodipine /Atorvastatin (Caduet®) Combination Tablets should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects intend to treat their cardiovascular disease who are prescribed Amlodipine /Atorvastatin (Caduet®) Combination Tablets by their Physicians

Exclusion Criteria:

Subjects who have been prescribed Amlodipine /Atorvastatin (Caduet®) Combination Tablets before.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects whom an investigator involving A3841063 prescribes the Amlodipine /Atorvastatin (Caduet®) Combination Tablets.
Sampling Method: Probability Sample
Enrollment: 1291 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841063&StudyName=Amlodipine/Atorvastatin%20%28Caduet%AE%29%20Drug%20Use%20Investigation%20%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 4, observational, open-label study conducted in Participants who were prescribed Amlodipine /Atorvastatin (Caduet®) Combination Tablets by their treating physician per usual clinical practice. Study drug was not provided by the Sponsor.
Groups:
- Amlodipine and Atorvastatin Combination Tablet: Participants who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Started | 1291
Completed | 1245
Not Completed | 46
Not completed — Protocol Violation | 46

BASELINE CHARACTERISTICS:
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 1245
Age, Customized [Number; unit: participants]
  <65 years | 377
  >=65 years | 868
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 787
  Male | 458
Type of Disease [Number; unit: participants]
  Hypertension | 1237
  Angina pectoris | 183
  Hypercholesterolemia | 1227
  Familial hypercholesterolemia | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in patients after administration of Caduet, irrespective of causal relationship to Caduet (including clinically problematic abnormal changes in laboratory test values). Treatment related Adverse Events were evaluated in company with the causal relationship to Caduet.
Time Frame: 8 weeks
Population: The safety analysis population consist of the cases that satisfy the participants conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 1245
participants | 18

2. Primary Outcome: Number of Participants That Responded to Amlodipine/Atorvastatin Treatment With Hypertension.
Description: The physician performed efficacy evaluations at the end of the observation period (or the time of discontinuing administration), compared with the data before the start of administration of this drug, and entered the results for Hypertension.
Time Frame: 8 weeks
Population: The efficacy analysis population basically consists of the evaluable cases with Hypertension in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 1202
participants | 1151

3. Primary Outcome: Number of Participants That Responded to Amlodipine/Atorvastatin Treatment With Angina Pectoris.
Description: The physician performed efficacy evaluations at the end of the observation period (or the time of discontinuing administration), compared with the data before the start of administration of this drug, and enteterd the results for Angina Pectoris.
Time Frame: 8 weeks
Population: The efficacy analysis population basically consists of the evaluable cases with Angina Pectoris in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 170
participants | 163

4. Primary Outcome: Number of Participants That Responded to Amlodipine/Atorvastatin Treatment With Hypercholesterolemia or Familial Hypercholesterolemia.
Description: The physician performed efficacy evaluations at the end of the observation period (or the time of discontinuing administration), compared with the data before the start of administration of this drug, and entered the results for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: The efficacy analysis population basically consists of the evaluable cases with Hypercholesterolemia or Familial Hypercholesterolemia in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 1057
participants | 1034

5. Secondary Outcome: Number of Treatment Related Unlisted Adverse Events in Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in patients after administration of Caduet, irrespective of causal relationship to Caduet (including clinically problematic abnormal changes in laboratory test values). Number of Treatment Related Adverse Events were evaluated in company with the causal relationship to Caduet. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: 8 weeks
Population: The safety analysis population consists of the cases that satisfy the participants conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Number analyzed (Participants) | 1245
participants
  Anaemia | 1
  Hypoproteinaemia | 1

6. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Gender.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether male or female is significant risk factor.
Time Frame: 8 weeks
Population: The safety analysis population consists of the cases that satisfy the cases conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Groups:
- Male: Male participants who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Female: Female participants who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 458 | 787
participants | 7 | 11
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "male and female" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.812, Fisher Exact

7. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Age.
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether <65 years or >=65 years is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- <65 Years: Participants with <65 years who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- >=65 Years: Participants with >=65 years who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 377 | 868
participants | 5 | 13
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is there is no difference between "<65 years and >=65 years" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

8. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Hypertension.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hypertension is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Without Hypertension: Participants without Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Hypertension: Participants with Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Hypertension | With Hypertension
Number analyzed (Participants) | 8 | 1237
participants | 0 | 18
Statistical Analysis 1: Comparison: Without Hypertension vs With Hypertension; The risk factor tested was "Hypertension". The null hypothesis is there is no difference between "with Hypetension and without Hypertension" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

9. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Hypertension Severity.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether Hypertension severity, "ClassⅠ, ClassⅡ, or ClassⅢ" is significant risk factor. Hypertension severity is defined by Guideline for the Management of hypertension (The Japan Society of Hypertension).
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- ClassⅠ: Participants with ClassⅠ Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- ClassⅡ: Participants with ClassⅡ Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- ClassⅢ: Participants with ClassⅢ Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | ClassⅠ | ClassⅡ | ClassⅢ
Number analyzed (Participants) | 656 | 351 | 95
participants | 5 | 4 | 3
Statistical Analysis 1: Comparison: ClassⅠ vs ClassⅡ vs ClassⅢ; The risk factor tested was "Hypertension severity". The null hypothesis is there is no difference among "ClassⅠHypertension, ClassⅡ Hypertension, and ClassⅢ Hypertension" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.112, Fisher Exact

10. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Angina Pectoris.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Angina pectoris is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Without Angina Pectoris: Participants without Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Angina Pectoris: Participants with Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Angina Pectoris | With Angina Pectoris
Number analyzed (Participants) | 1062 | 183
participants | 18 | 0
Statistical Analysis 1: Comparison: Without Angina Pectoris vs With Angina Pectoris; The risk factor tested was "Angina Pectoris". The null hypothesis is there is no difference between "with Angina Pectoris and without Angina Pectoris" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.093, Fisher Exact

11. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Hypercholesterolemia.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hypercholesterolemia is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Without Hypercholesterolemia: Participants without Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Hypercholesterolemia: Participants with Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Hypercholesterolemia | With Hypercholesterolemia
Number analyzed (Participants) | 18 | 1227
participants | 0 | 18
Statistical Analysis 1: Comparison: Without Hypercholesterolemia vs With Hypercholesterolemia; The risk factor tested was "Hypercholesterolemia". The null hypothesis is there is no difference between "with Hypercholesterolemia and without Hypercholesterolemia" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

12. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Hypercholesterolemia Expression Type.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether Hypercholesterolemia expression type, "Ⅰ, Ⅱa, Ⅱb, Ⅲ, Ⅳ, or Ⅴ" is significant risk factor. Hypercholesterolemia expression types are defined by Japan Atherosclerosis Society Guideline for Prevention of Atherosclerosis Cardiovascular Diseases.
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Type Ⅰ: Participants with expression type Ⅰ Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅱa: Participants with expression type Ⅱa Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅱb: Participants with expression type Ⅱb Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅲ: Participants with expression type Ⅲ Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅳ: Participants with expression type Ⅳ Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅴ: Participants with expression type Ⅴ Hypercholesterolemia who took Amlodipine /Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Type Ⅰ | Type Ⅱa | Type Ⅱb | Type Ⅲ | Type Ⅳ | Type Ⅴ
Number analyzed (Participants) | 15 | 609 | 207 | 12 | 6 | 0
participants | 0 | 10 | 2 | 0 | 0 |
Statistical Analysis 1: Comparison: Type Ⅰ vs Type Ⅱa vs Type Ⅱb vs Type Ⅲ vs Type Ⅳ vs Type Ⅴ; The risk factor tested was "Hypercholesterolemia expression type". The null hypothesis is there is no difference among "expression type Ⅰ, expression type Ⅱa, expression type Ⅱb, expression type Ⅲ, expression type, expression type Ⅳ, and expression type Ⅴ" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.839, Fisher Exact

13. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Familial Hypercholesterolemia.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Familial Hypercholesterolemia is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- Without Familial Hypercholesterolemia: Participants without Familial Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Familial Hypercholesterolemia: Participants with Familial Hypercholesterolemia who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Familial Hypercholesterolemia | With Familial Hypercholesterolemia
Number analyzed (Participants) | 1231 | 14
participants | 18 | 0
Statistical Analysis 1: Comparison: Without Familial Hypercholesterolemia vs With Familial Hypercholesterolemia; The risk factor tested was "Familial Hypercholesterolemia". The null hypothesis is there is no difference between "with Familial Hypercholesterolemia and without Familial Hypercholesterolemia" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

14. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Hepatic Dysfunction.
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hepatic Dysfunction is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- Without Hepatic Dysfunction: Participants without Hepatic Dysfunction who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Hepatic Dysfunction: Participants with Hepatic Dysfunction who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Hepatic Dysfunction | With Hepatic Dysfunction
Number analyzed (Participants) | 1087 | 145
participants | 14 | 2
Statistical Analysis 1: Comparison: Without Hepatic Dysfunction vs With Hepatic Dysfunction; The risk factor tested was "Hepatic Dysfunction". The null hypothesis is there is no difference between "with Hepatic Dysfunction and without Hepatic Dysfunction" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 1.000, Fisher Exact

15. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Renal Dysfunction.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Renal Dysfunction is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- Without Renal Dysfunction: Participants without Renal Dysfunction who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Renal Dysfunction: Participants with Renal Dysfunction who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Renal Dysfunction | With Renal Dysfunction
Number analyzed (Participants) | 1123 | 108
participants | 14 | 2
Statistical Analysis 1: Comparison: Without Renal Dysfunction vs With Renal Dysfunction; The risk factor tested was "Renal Dysfunction". The null hypothesis is there is no difference between "with Renal Dysfunction and without Renal Dysfunction" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.644, Fisher Exact

16. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Complications.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Complications is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- Without Complications: Participants without Complications who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Complications: Participants with Complications who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Complications | With Complications
Number analyzed (Participants) | 568 | 677
participants | 5 | 13
Statistical Analysis 1: Comparison: Without Complications vs With Complications; The risk factor tested was "Complications". The null hypothesis is there is no difference between "with Complications and without Complications" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.155, Fisher Exact

17. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets -Concomitant Drugs.
Description: Number of participants with Treatment Related Adverse Events(TRAEs) of Amlodipine/Atorvastatin Combination Tablets to determine whether Concomitant Drugs is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Groups:
- Without Concomitant Drugs: Participants without Concomitant Drugs who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- With Concomitant Drugs: Participants with Concomitant Drugs who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Without Concomitant Drugs | With Concomitant Drugs
Number analyzed (Participants) | 360 | 885
participants | 3 | 15
Statistical Analysis 1: Comparison: Without Concomitant Drugs vs With Concomitant Drugs; The risk factor tested was "Concomitant Drugs". The null hypothesis is there is no difference between "with Concomitant Drugs and without Concomitant Drugs" in the Incidence Rate of Treatment Related Adverse Events(TRAEs); Test type: Superiority or Other; p = 0.305, Fisher Exact

18. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Gender.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether male or female is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Male: Male Participants who took Amlodipine /Atorvastatin Combination Tablets according to Japanese Package Insert.
- Female: Female Participants who took Amlodipine /Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 438 | 764
participants | 415 | 736
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "males and females" in the participants of responders; Test type: Superiority or Other; p = 0.234, Fisher Exact

19. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Age.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether <65 years or >=65 is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 365 | 837
participants | 347 | 804
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is there is no difference between "<65 years and >=65 years" in the participants of responders; Test type: Superiority or Other; p = 0.439, Fisher Exact

20. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Hypertension Severity.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether Hypertension severity, "ClassⅠ, ClassⅡ, or ClassⅢ" is significant risk factor for Hypertension. Hypertension severity is defined by Guideline for the Management of hypertension (The Japan Society of Hypertension).
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- ClassⅡ: Participants with ClassⅡ Hypertension who took Amlodipine /Atorvastatin Combination Tablets according to Japanese Package Insert.
- ClassⅢ: Participants with Class Ⅲ Hypertension who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | ClassⅠ | ClassⅡ | ClassⅢ
Number analyzed (Participants) | 644 | 339 | 90
participants | 615 | 325 | 85
Statistical Analysis 1: Comparison: ClassⅠ vs ClassⅡ vs ClassⅢ; The risk factor tested was "Hypertension severity". The null hypothesis is there is no difference among "ClassⅠHypertension, ClassⅡ Hypertension, and ClassⅢ Hypertension" in the participants of responders; Test type: Superiority or Other; p = 0.761, Fisher Exact

21. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Hepatic Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hepatic Dysfunction is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Without Hepatic Dysfunction | With Hepatic Dysfunction
Number analyzed (Participants) | 1053 | 137
participants | 1008 | 131
Statistical Analysis 1: Comparison: Without Hepatic Dysfunction vs With Hepatic Dysfunction; The risk factor tested was "Hepatic Dysfunction". The null hypothesis is there is no difference between "with and without Hepatic Dysfunction" in the participants of responders; Test type: Superiority or Other; p = 1.000, Fisher Exact

22. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Renal Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Renal Dysfunction is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Without Renal Dysfunction | With Renal Dysfunction
Number analyzed (Participants) | 1085 | 104
participants | 1036 | 102
Statistical Analysis 1: Comparison: Without Renal Dysfunction vs With Renal Dysfunction; The risk factor tested was "Renal Dysfunction". The null hypothesis is there is no difference between "with and without Renal Dysfunction" in the participants of responders; Test type: Superiority or Other; p = 0.310, Fisher Exact

23. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Complications.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Complications is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Without Complications | With Complications
Number analyzed (Participants) | 555 | 647
participants | 527 | 624
Statistical Analysis 1: Comparison: Without Complications vs With Complications; The risk factor tested was "Complications". The null hypothesis is there is no difference between "with and without Complications" in the participants of responders; Test type: Superiority or Other; p = 0.251, Fisher Exact

24. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypertension -Concomitant Drugs.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Concomitant Drugs is significant risk factor for Hypertension.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Without Concomitant Drugs | With Concomitant Drugs
Number analyzed (Participants) | 355 | 847
participants | 339 | 812
Statistical Analysis 1: Comparison: Without Concomitant Drugs vs With Concomitant Drugs; The risk factor tested was "Concomitant Drugs". The null hypothesis is there is no difference between "with and without Concomitant Drugs" in the participants of responders; Test type: Superiority or Other; p = 0.756, Fisher Exact

25. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Gender.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether male or female is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Male | Female
Number analyzed (Participants) | 79 | 91
participants | 75 | 88
Statistical Analysis 1: Comparison: Male vs Female; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.706, Fisher Exact

26. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Age.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether <65 years or >=65 is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 45 | 125
participants | 45 | 118
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.192, Fisher Exact

27. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Angina Pectoris Severity.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether Angina Pectoris functional classification Severity, "Class1, Class2, Class3, or Class4" is significant risk factor for Angina Pectoris. Angina Pectoris functional classification Severity is defined by Canadian Cardiovascular Society functional Classification of Angina.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Class1: Participants with Class1 Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Class2: Participants with Class2 Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Class3: Participants with Class3 Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Class4: Participants with Class4 Angina Pectoris who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Class1 | Class2 | Class3 | Class4
Number analyzed (Participants) | 125 | 14 | 2 | 2
participants | 122 | 11 | 2 | 1
Statistical Analysis 1: Comparison: Class1 vs Class2 vs Class3 vs Class4; The risk factor tested was "Angina Pectoris Severity". The null hypothesis is there is no difference among "Class1, Class2, Class3, and Class4" in the participants of responders; Test type: Superiority or Other; p = 0.005, Fisher Exact

28. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Hepatic Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hepatic Dysfunction is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Without Hepatic Dysfunction | With Hepatic Dysfunction
Number analyzed (Participants) | 152 | 18
participants | 145 | 18
Statistical Analysis 1: Comparison: Without Hepatic Dysfunction vs With Hepatic Dysfunction; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 1.000, Fisher Exact

29. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Renal Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Renal Dysfunction is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Without Renal Dysfunction | With Renal Dysfunction
Number analyzed (Participants) | 144 | 25
participants | 137 | 25
Statistical Analysis 1: Comparison: Without Renal Dysfunction vs With Renal Dysfunction; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.596, Fisher Exact

30. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Complications.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Angina Pectoris is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Without Complications | With Complications
Number analyzed (Participants) | 61 | 109
participants | 57 | 106
Statistical Analysis 1: Comparison: Without Complications vs With Complications; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.252, Fisher Exact

31. Secondary Outcome: Risk Factors for the Proportion of Responders for Angina Pectoris -Concomitant Drugs.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Concomitant Drugs is significant risk factor for Angina Pectoris.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Without Concomitant Drugs | With Concomitant Drugs
Number analyzed (Participants) | 23 | 147
participants | 22 | 141
Statistical Analysis 1: Comparison: Without Concomitant Drugs vs With Concomitant Drugs; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 1.000, Fisher Exact

32. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Gender.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether male or female is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Male | Female
Number analyzed (Participants) | 390 | 667
participants | 380 | 654
Statistical Analysis 1: Comparison: Male vs Female; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.518, Fisher Exact

33. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Age.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether <65 years or >=65 is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 313 | 744
participants | 305 | 729
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.645, Fisher Exact

34. Secondary Outcome: Risk Factor for the Proportion of Responders of Amlodipine/Atorvastatin Combination Tablets for Hypercholesterolemia or Familial Hypercholesterolemia - Hypercholesterolemia Expression Type.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether Hypercholesterolemia expression type, "Ⅰ, Ⅱa, Ⅱb, Ⅲ, Ⅳ, or Ⅴ" is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia. Hypercholesterolemia expression types are defined by Japan Atherosclerosis Society Guideline for Prevention of Atherosclerosis Cardiovascular Diseases.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Type Ⅰ: Participants with expression type Ⅰ who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅱa: Participants with expression type Ⅱa who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅱb: Participants with expression type Ⅱb who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅲ: Participants with expression type Ⅲ who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅳ: Participants with expression type Ⅳ who took Amlodipine/Atorvastatin Combination Tablets according to Japanese Package Insert.
- Type Ⅴ: Participants with expression type Ⅴ who took Amlodipine /Atorvastatin Combination Tablets according to Japanese Package Insert.
Arm/Group | Type Ⅰ | Type Ⅱa | Type Ⅱb | Type Ⅲ | Type Ⅳ | Type Ⅴ
Number analyzed (Participants) | 13 | 541 | 187 | 11 | 5 | 0
participants | 13 | 533 | 180 | 10 | 5 |
Statistical Analysis 1: Comparison: Type Ⅰ vs Type Ⅱa vs Type Ⅱb vs Type Ⅲ vs Type Ⅳ vs Type Ⅴ; The risk factor tested was "Hypercholesterolemia expression type". The null hypothesis is there is no difference among "expression type Ⅰ, expression type Ⅱa, expression type Ⅱb, expression type Ⅲ, expression type, expression type Ⅳ, and expression type Ⅴ" in the participants of responders; Test type: Superiority or Other; p = 0.130, Fisher Exact

35. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Hepatic Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Hepatic Dysfunction is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Without Hepatic Dysfunction | With Hepatic Dysfunction
Number analyzed (Participants) | 922 | 127
participants | 904 | 122
Statistical Analysis 1: Comparison: Without Hepatic Dysfunction vs With Hepatic Dysfunction; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.185, Fisher Exact

36. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Renal Dysfunction.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Renal Dysfunction is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Without Renal Dysfunction | With Renal Dysfunction
Number analyzed (Participants) | 959 | 89
participants | 937 | 88
Statistical Analysis 1: Comparison: Without Renal Dysfunction vs With Renal Dysfunction; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.714, Fisher Exact

37. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Complications.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Complications is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Without Complications | With Complications
Number analyzed (Participants) | 492 | 565
participants | 482 | 552
Statistical Analysis 1: Comparison: Without Complications vs With Complications; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; p = 0.835, Fisher Exact

38. Secondary Outcome: Risk Factors for the Proportion of Responders for Hypercholesterolemia or Familial Hypercholesterolemia -Concomitant Drugs.
Description: Number of Participants with responders of Amlodipine/Atorvastatin Combination Tablets to determine whether with or without Concomitant Drugs is significant risk factor for Hypercholesterolemia or Familial Hypercholesterolemia.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Without Concomitant Drugs | With Concomitant Drugs
Number analyzed (Participants) | 310 | 747
participants | 306 | 728
Statistical Analysis 1: Comparison: Without Concomitant Drugs vs With Concomitant Drugs; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.252, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Amlodipine and Atorvastatin Combination Tablet
Serious Adverse Events (participants affected / at risk) | 1/1245
Other Adverse Events (participants affected / at risk) | 17/1245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine and Atorvastatin Combination Tablet (N=1245)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine and Atorvastatin Combination Tablet (N=1245)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3)
Blood glucose increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.